CLINICAL TRIAL: NCT04762784
Title: A Prospective, Controlled, Interventional Study to Evaluate the Efficacy and Safety of Tocilizumab in the Treatment of Idiopathic Retroperitoneal Fibrosis
Brief Title: A Prospective Study of Tocilizumab in the Treatment of Idiopathic Retroperitoneal Fibrosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wen Zhang, Professor, Peking Union Medical College Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: tocilizumab treatment for IRPF
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Idiopathic Retroperitoneal Fibrosis
Keywords: idiopathic retroperitoneal fibrosis; Tocilizumab; Response
MeSH Terms: conditions — Retroperitoneal Fibrosis | interventions — tocilizumab; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab treatment (Experimental): Tocilizumab is a recombinant humanized monoclonal antibody against human interleukin-6 (IL-6) receptor. Tocilizumab acts by inhibiting the activity of IL-6 receptor. IL-6 is a pro-inflammatory cytokine whose release can trigger a series of downstream pro-inflammatory responses. Tocilizumab inhibits IL-6 signal transduction by blocking the binding of IL-6 to soluble and membrane-bound IL-6 receptors, thereby reducing pathological inflammatory responses.
  Interventions: Drug: Tocilizumab
- Glucocorticoids monotherapy (Active Comparator): Glucocorticoids has fast onset of action and multiple anti-inflammatory effects.The conventional protocol is oral prednisone, followed by a slow tapering over 4 weeks. Besides, precautionary measures need to be taken against possible complications brought by the application of corticosteroids such as infections, diabetes mellitus, hypertension, Cushing's syndrome and osteoporosis, etc.
  Interventions: Drug: Glucocorticoids

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab treatment: Tocilizumab infusion 8mg/Kg，Once per month for 3 months.
  Arms: Tocilizumab treatment
Drug: Glucocorticoids — Prednisone/prednisolone: started at 0.6-0. 8mg/kg.d for 2 to 4 weeks, tapered at 5mg per 1-2 weeks to equal to or less than 15mg per day in 3 months.
  Arms: Glucocorticoids monotherapy

SUMMARY:
This is a prospective study to investigate the treatment response of Tocilizumab on patients with idiopathic retroperitoneal fibrosis（IRPF）.

Methods: All the patients fulfilling diagnostic criteria of IRPF would be enrolled. The IRPF patients will accept Tocilizumab or Glucocorticoid monotherapy for 3 months.

Endpoints: The primary endpoint is to investigate the response of Tocilizumab on IRPF patients; the secondary endpoints include the decrease of inflammatory markers, side effect.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 diagnosed as IRPF: The diagnosis of idiopathic retroperitoneal fibrosis is based on the following aspects :(1) the swelling of retroperitoneal tissue , which seems neoplastic; (2) A large number of lymphocytes proliferated and infiltrated in the affected tissues and organs, and tissues showed inflammation, fibrosis and sclerosis, in which IgG4-positive cells accounted for less than 50% of plasma cells; (3) Increased inflammatory markers, such as ESR and CRP; (4) Good response to glucocorticoid therapy.

Exclusion Criteria:

* malignancy retroperitoneal fibrosis secondary to other diseases or drug treatment or abdominal surgeries.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-02-10 (Estimated); Study Completion 2023-02-10 (Estimated)

PRIMARY OUTCOMES:
remission | 5 years
  Remission is achieved when symptoms are alleviated and laboratory tests return to normal levels or radiologic improvement is observed.

SECONDARY OUTCOMES:
relapse | 5 years
  Participants have recurrence of symptoms and laboratory abnormalities.

OTHER OUTCOMES:
adverse events | 5 years
  Participants suffer from adverse events due to the drug treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marzano A, Trapani A, Leone N, Actis GC, Rizzetto M. Treatment of idiopathic retroperitoneal fibrosis using cyclosporin. Ann Rheum Dis. 2001 Apr;60(4):427-8. doi: 10.1136/ard.60.4.427. PMID 11247880
- [Background] Schultz O, Schuchmann S, Burmester GR, Buttgereit F. Case number 26: systemic idiopathic fibrosis associated with aortitis. Ann Rheum Dis. 2003 May;62(5):486. doi: 10.1136/ard.62.5.486. No abstract available. PMID 12695167
- [Background] Summaries for patients. Tamoxifen for the treatment of retroperitoneal fibrosis. Ann Intern Med. 2006 Jan 17;144(2):I51. doi: 10.7326/0003-4819-144-2-200601170-00002. No abstract available. PMID 16418405
- [Background] van Bommel EF, Hendriksz TR, Huiskes AW, Zeegers AG. Brief communication: tamoxifen therapy for nonmalignant retroperitoneal fibrosis. Ann Intern Med. 2006 Jan 17;144(2):101-6. doi: 10.7326/0003-4819-144-2-200601170-00007. PMID 16418409
- [Background] Vaglio A, Salvarani C, Buzio C. Retroperitoneal fibrosis. Lancet. 2006 Jan 21;367(9506):241-51. doi: 10.1016/S0140-6736(06)68035-5. PMID 16427494
- [Background] Vaglio A, Greco P, Buzio C. Tamoxifen therapy for retroperitoneal fibrosis. Ann Intern Med. 2006 Apr 18;144(8):619; author reply 619-20. doi: 10.7326/0003-4819-144-8-200604180-00017. No abstract available. PMID 16618960
- [Background] Jagadesham VP, Scott DJ, Carding SR. Abdominal aortic aneurysms: an autoimmune disease? Trends Mol Med. 2008 Dec;14(12):522-9. doi: 10.1016/j.molmed.2008.09.008. Epub 2008 Nov 6. PMID 18980864
- [Background] Qian Q, Kashani KB, Miller DV. Ruptured abdominal aortic aneurysm related to IgG4 periaortitis. N Engl J Med. 2009 Sep 10;361(11):1121-3. doi: 10.1056/NEJMc0905265. No abstract available. PMID 19741239
- [Background] Scheel PJ Jr, Feeley N, Sozio SM. Combined prednisone and mycophenolate mofetil treatment for retroperitoneal fibrosis: a case series. Ann Intern Med. 2011 Jan 4;154(1):31-6. doi: 10.7326/0003-4819-154-1-201101040-00005. PMID 21200036
- [Background] Swartz R, Scheel P. Retroperitoneal fibrosis: gaining traction on an enigma. Lancet. 2011 Jul 23;378(9788):294-6. doi: 10.1016/S0140-6736(11)60880-5. Epub 2011 Jul 4. No abstract available. PMID 21733569
- [Background] Vaglio A, Palmisano A, Alberici F, Maggiore U, Ferretti S, Cobelli R, Ferrozzi F, Corradi D, Salvarani C, Buzio C. Prednisone versus tamoxifen in patients with idiopathic retroperitoneal fibrosis: an open-label randomised controlled trial. Lancet. 2011 Jul 23;378(9788):338-46. doi: 10.1016/S0140-6736(11)60934-3. Epub 2011 Jul 4. PMID 21733570
- [Background] Binder M, Uhl M, Wiech T, Kollert F, Thiel J, Sass JO, Walker UA, Peter HH, Warnatz K. Cyclophosphamide is a highly effective and safe induction therapy in chronic periaortitis: a long-term follow-up of 35 patients with chronic periaortitis. Ann Rheum Dis. 2012 Feb;71(2):311-2. doi: 10.1136/annrheumdis-2011-200148. Epub 2011 Aug 22. No abstract available. PMID 21859695